CLINICAL TRIAL: NCT01191190
Title: A Phase II Study of Ofatumumab in Combination With High-dose Methylprednisolone in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Ofatumumab and High-dose Methylprednisolone in Patients With Chronic Lymphocytic Leukemia (CLL)
Acronym: CRC027
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Januario Castro, M.D. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Januario Castro, M.D., Principal Investigator, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100429
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: CLL
Keywords: Leukemia; Chronic leukemia; Chronic Lymphocytic Leukemia; Relapsed; Refractory
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab/HDMP (Experimental): High dose methylprednisolone sodium succinate (HDMP) at 1gm/m2 daily as infusion for 3 consecutive days every cycle.
  Ofatumumab 300mg administered Day1 of cycle 1 followed by 12 doses of 1000mg administered.
  Each patient may receive 3 cycles of treatment in the absence of progressive disease or significant toxicity.
  Interventions: Drug: Ofatumumab/HDMP

INTERVENTIONS:
Drug: Ofatumumab/HDMP — High dose methylprednisolone sodium succinate (HDMP) at 1gm/m2 daily as infusion for 3 consecutive days every cycle.
  Ofatumumab 300mg administered Day1 of cycle 1 followed by 12 doses of 1000mg administered based on specific schedule.
  Each patient will receive a maximum of 3 cycles (one cycle is 28 days)
  Other Names: Arzerra; HuMax-CD20

SUMMARY:
Patients who have relapsed/refractory CLL and require therapy as per iwCLL guidelines will be eligible. Subjects will receive a treatment with ofatumumab and HDMP for three consecutive 4 week cycles. The primary endpoint is to determine the complete response (CR) to therapy and the secondary endpoints will assess the safety and tolerability of the regimen, the impact of the treatment on progression free, treatment free, overall survival, and pharmacokinetics of ofatumumab. Patients will receive allopurinol for tumor-lysis prophylaxis and antimicrobial prophylaxis.

DETAILED DESCRIPTION:
Patients who have relapsed/refractory CLL and require therapy as per iwCLL guidelines will be eligible. Subjects will receive a treatment with ofatumumab and HDMP for three consecutive 4 week cycles. The primary endpoint is to determine the complete response (CR) to therapy and the secondary endpoints will assess the safety and tolerability of the regimen, the impact of the treatment on progression free, treatment free, overall survival, and pharmacokinetics of ofatumumab. Cycles 1-3 will be administered without scheduled interruption every 28 days for a total of 12 weeks of therapy. Patients will receive allopurinol for tumor-lysis prophylaxis and antimicrobial prophylaxis. Blood glucose levels will be monitored immediately after HDMP infusion by finger stick glucometry. Two months following completion of treatment a response assessment will occur per iwCLL guidelines. The treatment will be administered as outpatient, and each cycle will be four weeks in duration.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated patients with a diagnosis of CLL
2. Previous treatment with any monoclonal antibody or chemotherapy regardless of response as defined by the iwCLL Working Group Guidelines as evidenced by:

   * progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
   * massive (i.e. at least 6cm below the left costal margin) or progressive or symptomatic splenomegaly
   * massive nodes (i.e. at least 10cm in longest diameter) or progressive or symptomatic lymphadenopathy.
   * progressive lymphocytosis with an increase of more than 50% over a 2-month period or lymphocyte doubling time (LDT) of less than 6 months.
   * autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy (See Section 10.2)
3. Constitutional symptoms, defined as any one or more of the following disease-related symptoms or signs: unintentional weight loss of 10% or more within the previous 6 months significant fatigue (i.e. ECOG PS 2 or worse, inability to work or perform usual activities), fevers higher than 100.5ºF or 38.0ºC for 2 or more weeks without other evidence of infection, night sweats for more than 1 month without evidence of infection
4. Subjects must be 18 years of age or older, male or female.
5. ECOG performance status of 0-2.
6. Subjects must be able to give informed consent.
7. Females of child bearing potential(FCBP)† must have a negative serum or urine pregnancy test within 10 - 14 days prior to and again within 24 hours of starting treatment and agree to use a medically accepted contraceptive method for the duration of this study.

Exclusion Criteria:

1. Hepatitis BsAg positive, Hepatitis BcAb positive, and Hepatitis C positive patients.
2. Known HIV positive patients.
3. Diabetics.
4. Patients with uncontrolled Autoimmune Hemolytic Anemia (AIHA) or autoimmune thrombocytopenia (ITP).
5. Screening laboratory values within these ranges: platelets <50 x 109/L, neutrophils <1.0 x 109/L, creatinine >2.0 times upper normal limit,total bilirubin >1.5 times upper normal limit (unless a known history of Gilbert's disease), ALT >2.5 times upper normal limit (unless due to disease involvement of liver), alkaline phosphatase >2.5 times upper normal limit (unless due to disease involvement of the liver or bone marrow)
6. Inability to provide informed consent.
7. Concurrent malignancy (excluding basal and squamous cell skin cancers).
8. Active fungal, bacterial, and/or viral infection.
9. History of peptic ulcer disease resulting in GI bleeding within the last 6 months.
10. Untreated metabolic disorders such as hypothyroidism and Cushing's disease.
11. History of steroid-induced psychosis.
12. Estimated life expectancy of less than 3 months by the investigator's best clinical judgment.
13. Serious medical condition that would render the subject medically unstable.
14. Women who are pregnant or breast-feeding.
15. History of Pancreatitis.
16. History of Diverticulitis.
17. Patients with known hypersensitivity to ofatumumab or known history of anaphylaxis to Rituximab or alemtuzumab.
18. Concurrent use of other anti-cancer agents or treatments.
19. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Januario Castro, MD, Principal Investigator — University of California, San Diego; Thomas J Kipps, MD, PhD, Principal Investigator — Director of the CLL Research Consortium and University of California San Diego
Locations (2):
- United States (2):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California San Diego, Moores Cancer Center, La Jolla, California

REFERENCES:
- [Background] Castro JE, James DF, Sandoval-Sus JD, Jain S, Bole J, Rassenti L, Kipps TJ. Rituximab in combination with high-dose methylprednisolone for the treatment of chronic lymphocytic leukemia. Leukemia. 2009 Oct;23(10):1779-89. doi: 10.1038/leu.2009.133. Epub 2009 Aug 20. PMID 19693094
- [Background] Castro JE, Sandoval-Sus JD, Bole J, Rassenti L, Kipps TJ. Rituximab in combination with high-dose methylprednisolone for the treatment of fludarabine refractory high-risk chronic lymphocytic leukemia. Leukemia. 2008 Nov;22(11):2048-53. doi: 10.1038/leu.2008.214. Epub 2008 Aug 28. PMID 18754025
- See also: Moore's UCSD Cancer Center — http://cancer.ucsd.edu/
- See also: Website for the Chronic Lymphocytic Leukemia Research Consortium — http://cllresearch.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab/HDMP: High dose methylprednisolone sodium succinate (HDMP) at 1gm/m2 daily as infusion for 3 consecutive days every cycle.
  Ofatumumab 300mg administered Day1 of cycle 1 followed by 12 doses of 1000mg administered.
  Each patient may receive 3 cycles of treatment in the absence of progressive disease or significant toxicity.
  Ofatumumab/HDMP: High dose methylprednisolone sodium succinate (HDMP) at 1gm/m2 daily as infusion for 3 consecutive days every cycle.
  Ofatumumab 300mg administered Day1 of cycle 1 followed by 12 doses of 1000mg administered based on specific schedule.
  Each patient will receive a maximum of 3 cycles (one cycle is 28 days)
Period: Overall Study
Arm/Group | Ofatumumab/HDMP
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: IwCLL-WG Defined Complete Response (CR)
Description: Responses were assessed two months after completion of therapy.
  Criteria for complete remission is assessed with: a bone marrow biopsy and repeat CT scan (abdominal, chest and pelvis if initial was abnormal) to confirm iwCLL-WG defined CR.
  iwCLL-WG Complete Response is defined as:
  * Peripheral blood lymphocytes (evaluated by blood and differential count) below 4 x 109/L (4000/L).
  * Absence of lymphadenopathy (>1.5 cm)of physical exam; AND
  * No hepatomegaly and splenomegaly on physical exam; AND
  * Absence of constitutional symptoms; AND
  * Normal complete blood count as exhibited by neutrophils ≥ 1,500/μl, platelets > 100,000/μl, hemoglobin > 11.0g/dL (non-transfused), and lymphocyte count < 5,000/μl; AND
  * Bone marrow aspirate and biopsy must be normocellular for age with <30% of nucleated cells being lymphocytes. Lymphoid nodules must be absent
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
participants | 1

2. Secondary Outcome: IwCLL-WG Defined Overall Response Rate (ORR)
Description: Responses were assessed two months after completion of therapy. Overall Response Rate (ORR) = CR + PR
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
participants | 17

3. Secondary Outcome: IwCLL-WG Defined Nodular Partial Response (PR)
Description: Responses were assessed two months after completion of therapy.
  Partial Response is defined as:
  * Greater than or equal to 50% decrease in blood absolute lymphocyte count from pre-treatment value; AND
  * Greater than or equal to 50% reduction in lymphadenopathy from pre-treatment value; AND
  * Greater than or equal to 50% reduction in splenomegaly/hepatomegaly from pre-treatment value.
  In addition, patients need to have at least ONE of the following:
  * Neutrophils ≥ 1,500/μl or ≥ 50% improvement from pre-treatment value; AND / OR
  * Platelets > 100,000/μl or 50% improvement from pre-treatment value; AND / OR
  * Hemoglobin > 11.0 gm/dl (non-transfused) or 50% improvement from pre-treatment value.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
participants | 2

4. Secondary Outcome: IwCLL-WG Defined Partial Response (PR)
Description: Responses were assessed two months after completion of therapy
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
participants | 14

5. Secondary Outcome: IwCLL-WG Defined Stable Disease (SD)
Description: Responses were assessed two months after completion of therapy.
  Subjects who do not fulfill the criteria for complete or partial response as defined above but do not exhibit progressive disease will be considered as having stable disease.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
participants | 3

6. Secondary Outcome: IwCLL-WG Defined Progressive Disease (PD)
Description: Responses were assessed two months after completion of therapy
  Progressive Disease is defined as:
  * Greater than or equal to 50% increase in the products of at least two lymph nodes on two consecutive determinations two weeks apart (at least one lymph node must be ≥ 2 cm; or the appearance of a new palpable lymph node; OR
  * Greater than or equal to 50% increase in the size of the liver and/or spleen as determined by measurement below the respective costal margins; or appearance of palpable hepatomegaly or splenomegaly, which was not previously present; OR
  * Greater than or equal to 50% increase in the absolute number of circulating lymphocytes to at least 5,000μl; OR
  * Transformation to a more aggressive histology (i.e., Richter's syndrome or prolymphocytic leukemia with ≥ 56% prolymphocytes);
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
participants | 1

7. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
months | 9.9 [2 to 34]

8. Secondary Outcome: Treatment-Free Survival
Time Frame: 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
months | 12.1 [2 to 36]

9. Secondary Outcome: Safety and Tolerability Measured Via Adverse Events
Description: Please see Adverse Event module for additional details.
Time Frame: 2 years
Population: Total number of participants who had at least 1 adverse event
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 21
participants | 21

10. Secondary Outcome: Detectable Minimal Residual Disease (MRD)
Description: The patient who achieved a CR did not have detectable MRD in the bone marrow by four-color flow cytometry (<0.1% of cells).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Ofatumumab/HDMP
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Arm/Group | Ofatumumab/HDMP
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab/HDMP (N=21)
Infusion reaction (Immune system disorders) | 11
Flushing (Immune system disorders) | 5
Allergic Reaction (Immune system disorders) | 1
Cough (General disorders) | 9
Edema (General disorders) | 7
Dizziness (General disorders) | 5
Hypotension (General disorders) | 4
Tachycardia (General disorders) | 4
Dyspnea (General disorders) | 4
Palpitations (General disorders) | 3
Arrythmia (General disorders) | 2
Non-ST elevation Myocardial Infarction (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 16
Pruritis (Skin and subcutaneous tissue disorders) | 11
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1
Atypical Squamous Proliferation, Folliculitis (Skin and subcutaneous tissue disorders) | 1
Lichenoid Dermatitis (Skin and subcutaneous tissue disorders) | 1
Elevated ALT (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 7
Elevated AST (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 4
Anorexia (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 2
Hyperbilirubinemia (Gastrointestinal disorders) | 1
Anemia (CTCAE) (Blood and lymphatic system disorders) | 18
Thrombocytopenia (CTCAE) (Blood and lymphatic system disorders) | 15
Neutropenia (CTCAE) (Blood and lymphatic system disorders) | 10
Leukocytopenia, not captured by neutropenia (Blood and lymphatic system disorders) | 2
Bleeding (superficial) (Blood and lymphatic system disorders) | 2
Upper Respiratory Infection (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Non-melanoma skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperglycemia (General disorders) | 18
Fatigue (General disorders) | 13
Hypocalcemia (General disorders) | 7
metabolic other Elevated LDH- (General disorders) | 7
Hypokalemia (General disorders) | 5
Diaphoresis (General disorders) | 4
Night Sweats (General disorders) | 4
Weight Gain (General disorders) | 4
Hypokalemia (General disorders) | 3
Weakness (General disorders) | 3
Fever (General disorders) | 3
Hypernatremia (General disorders) | 3
Hyperuricemia (General disorders) | 3
Weight Loss (General disorders) | 3
Rigors/ chills (General disorders) | 2
Hyperkalemia (General disorders) | 1
Insomnia (General disorders) | 15
Anxiety (General disorders) | 7
Paraethesias (General disorders) | 5
Headache (General disorders) | 4
Tremor (General disorders) | 3
Visual change (General disorders) | 2
Neuropathy (General disorders) | 2
Agitation (General disorders) | 2
Pharyngolaryngeal pain/itching (General disorders) | 4
Rhinnorhea (General disorders) | 4
Allergic rhinitis (General disorders) | 3
Dysguesia (General disorders) | 3
Weak Voice (General disorders) | 2
Dysphagia (General disorders) | 1
Oral ulcers (General disorders) | 1
Abdominal Pain (General disorders) | 5
Myalgia (General disorders) | 2
Lower Back Pain (General disorders) | 2
Creatinine elevation (Renal and urinary disorders) | 8
Kidney stones (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Penile blister (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes